CLINICAL TRIAL: NCT04084912
Title: The Effect of Preoperative Steroids Injection on Pain and Oedema After Total Knee Arthroplasty . A Double -Blinded Randomized Controlled Study.
Brief Title: Effect of Preoperative Steroid in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, DNKameel, physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: steroid injection in TKA
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Arthropathy of Knee
MeSH Terms: interventions — dexamethasone 21-phosphate; Steroids; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone group (Active Comparator): this group will receive one ampoule Intravenous injection of Dexamethasone Sodium Phosphate 2 ml . 8 mg once by the anesthesiologist immediately before skin incision
  Interventions: Drug: Dexamethasone Sodium Phosphate
- Placebo group (Placebo Comparator): this group will receive one ampoule Intravenous injection of Saline once by the anesthesiologist immediately before skin incision
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate — intravenous injection of one ampoule dexamethasone Sodium phosphate 2 ml 8 mg
  Other Names: Steroid
  Arms: Dexamethasone group
Drug: Saline Solution — intravenous injection of one ampoule saline
  Other Names: saline
  Arms: Placebo group

SUMMARY:
Detect the effect of preoperative steroid injection in total knee arthroplasty on post operative:

1. pain
2. oedema
3. nausea and vomiting
4. quadriceps power
5. knee flexion
6. wound complications

DETAILED DESCRIPTION:
Total knee arthroplasty has been identified as one of the most effective surgeries for knee arthritis. Many patients experience moderate to severe pain during the early postoperative period, as the surgery involves extensive bone resection and postsurgical serum levels of cytokine interleukin-6 and C-reactive protein may be elevated.Furthermore, many patients suffer postoperative nausea and vomiting after total knee arthroplasty . The inflammatory response after TKA is pronounced and a result of cumulative effects of anaesthesia and mechanical stress . Inadequate management of postoperative pain is relevant with a series of undesirable effects, including progression to a persistent pain, delayed functional recovery, increased the economic burden and patient dissatisfaction. Steroids may be associated with decreased levels of interleukin-6 and C reactive protein and may, thus, relieve the pain associated with surgery. Dexamethasone is a long-acting glucocorticoid that has been reported to inhibit peripheral phospholipase A, which decreases the pain-aggravating agents from the cyclooxygenase and lipoxygenase pathways . In addition, it reduces postoperative nausea and vomiting by exerting a central antiemetic effect by inhibiting prostaglandin synthesis and the release of endogenous opioids[5] . Some studies also reported potential adverse events, such as infection .

ELIGIBILITY:
Inclusion Criteria:

1. Any patient scheduled for primary total knee replacement arthroplasty

Exclusion Criteria:

1. Diabetic patients
2. Rheumatoid arthritis patients
3. Patients on regular steroid therapy
4. Patients refused to be enrolled in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain summarized in the first 14 days | 14 days
  postoperative pain summarized over first 14 days after surgery , assessed by a summation of Visual Analog Scale (VAS)-scores at day 1 , day 2 , day 3 and day 14 after surgery pain is monitored by Visual Analog Scale (VAS) 0-100 mm, where 0 is no pain and 100 is the worst pain one can imagine Moderate pain is considered a VAS >30 mm.

SECONDARY OUTCOMES:
Postoperative Thigh circumference in the first 14 days | 14 days
  Postoperative oedema will be assessed for all participants by measuring Thigh circumference 1 cm above the upper pole of the patella postoperatively at day 1,2,3 and 14
postoperative nausea and vomiting in the first 14 days | 14 days
  postoperative nausea and vomiting summarized over first 14 days after surgery , assessed by a summation of Visual Analog Scale (VAS)-scores at day 1 , day 2 , day 3 and day 14 after surgery Nausea and vomiting is monitored by Visual Analog Scale (VAS) 0-100 mm, where 0 is no nausea nor vomiting and 100 is the worst nausea and vomiting one can imagine Moderate pain is considered a VAS >30 mm.
postoperative knee flexion in the first 14 days | 14 days
  Knee flexion assessed over first 14 days after surgery assessed by knee range of motion measured by goniometer where straight knee joint measure 0 degree.
Surgical wound infection in the first 14 days | 14 days
  wound complications like infection to be reported: redness, discharge, infection, dehiscence, delayed healing (up to 2 wks) postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Bakr, asst. prof, Study Chair — Assiut University

REFERENCES:
- [Background] Xing LZ, Li L, Zhang LJ. Can intravenous steroid administration reduce postoperative pain scores following total knee arthroplasty?: A meta-analysis. Medicine (Baltimore). 2017 Jun;96(24):e7134. doi: 10.1097/MD.0000000000007134. PMID 28614237
- [Background] Rytter S, Stilling M, Munk S, Hansen TB. Methylprednisolone reduces pain and decreases knee swelling in the first 24 h after fast-track unicompartmental knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Jan;25(1):284-290. doi: 10.1007/s00167-014-3501-8. Epub 2015 Jan 7. PMID 25564196
- [Background] Fan Z, Ma J, Kuang M, Zhang L, Han B, Yang B, Wang Y, Ma X. The efficacy of dexamethasone reducing postoperative pain and emesis after total knee arthroplasty: A systematic review and meta-analysis. Int J Surg. 2018 Apr;52:149-155. doi: 10.1016/j.ijsu.2018.02.043. Epub 2018 Feb 23. PMID 29481989
- [Background] Meng J, Li L. The efficiency and safety of dexamethasone for pain control in total joint arthroplasty: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2017 Jun;96(24):e7126. doi: 10.1097/MD.0000000000007126. PMID 28614232
- [Background] Yue C, Wei R, Liu Y. Perioperative systemic steroid for rapid recovery in total knee and hip arthroplasty: a systematic review and meta-analysis of randomized trials. J Orthop Surg Res. 2017 Jun 27;12(1):100. doi: 10.1186/s13018-017-0601-4. PMID 28655354